CLINICAL TRIAL: NCT07385183
Title: CARE: Comprehensive Assessment of Real-world Effectiveness of F/TAF in Persons Who Use Drugs (PWUD)
Acronym: CARE
Status: Not yet recruiting | Type: Observational
Sponsor: Heather Henderson (Other)
Collaborators: Gilead Sciences (Industry); Tampa General Hospital (Other); University of South Florida (Other)
Responsible Party: Sponsor-Investigator, Heather Henderson, Assistant Professor, Emergency Medicine Director, Division of Social Emergency Medicine, Population and Global Health Program Director, Idea Exchange Tampa, University of South Florida
Organization: University of South Florida (Other)
Other Study IDs: CARE
Record Dates: First submitted 2026-01-06; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: People Who Inject Drugs; PrEP Adherence
Keywords: PrEP; People who Use/Inject Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PrEP arm: patients receiving PrEP and being followed for 1 year
  Interventions: Other: PrEP adherence; Other: PrEP perspectives
- Interview only group: patients who do not wish to receive PrEP and complete a single interview assessing why they do not want PrEP
  Interventions: Other: PrEP perspectives
- Clinician Interview: Collection clinician perceptions on PrEP
  Interventions: Other: PrEP perspectives

INTERVENTIONS:
Other: PrEP adherence — PrEP adherence: Determine adherence rates and persistence with PrEP regimen over time and understand the facilitators and barriers to adherence and persistence
  Groups: PrEP arm
Other: PrEP perspectives — Awareness and understanding of PrEP from non-PrEP using patients and clinicians who provide care for PWID.

SUMMARY:
This study looks at how to help people who use drugs start and keep taking medicine that can prevent HIV. The medicine is called PrEP (pre-exposure prophylaxis). The study investigators will use a pill called Descovy (F/TAF), which is already approved by the FDA for HIV prevention.

People who come to the emergency department (ED) and test negative for HIV may join the study. Some participants will start taking PrEP and will be followed for one year. Other participants will only do an interview about their thoughts on PrEP. The study investigators will also talk to doctors and peer support workers in the ED to learn what makes it easier or harder to offer PrEP.

The main goal is to see how well PrEP can be started and continued for people who use drugs. The study investigators will look at how many people start PrEP, how many keep taking it, and what helps or makes it hard to stay on PrEP. The study investigators will also learn about the best ways to connect people to care after they leave the ED.

This study does not test if the medicine works to prevent HIV-that is already known. Instead, it looks at real-life challenges and solutions for using PrEP in this group. The study may help improve HIV prevention and health care for people who use drugs.

ELIGIBILITY:
Inclusion Criteria:

* Prep Initiation Inclusion: 18 years of age or older; Communicate in English; Confirmatory test of HIV-negative; Documented or identified history of injection drug use within the last six-months or have documented or identified general drug use within the last twelve months; Be able to provide at least one contact person including name and phone number where participant can be reached for follow-up
* Clinician Interview Inclusion: At least 18 years of age; Healthcare provider or peer navigator, a person with lived experience in substance use disorder who will help navigate the patient through care, currently employed in TGH ED
* Interview Inclusion: At least 18 years of age; Communicate in English; Confirmatory test of HIV-negative; Documented or identified history of injection drug use within the last six-months or have documented or identified general drug use within the last twelve months;

Exclusion Criteria:

* PrEP Initiation Exclusion: Under 18 years of age; Determined to be HIV-positive following confirmatory testing; Have a CrCl of less than 30ml/min, making them only eligible for long-acting injectable PrEP if CrCl is a limiting factor for oral PrEP; Have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent; Are currently incarcerated or have pending legal action that may prevent an individual from completing the study; Pregnant.
* Clinician Interview Exclusion: Under 18 years of age; Not currently employed as a healthcare provider or peer navigator in the TGH ED.
* Interview Exclusion: Under 18 years of age; Have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent; Are currently incarcerated or have pending legal action that may prevent an individual from completing the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tampa General Hospital Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adherence and Persistence Rates of Oral PrEP (F/TAF) Among Persons Who Use Drugs Over 12 Months | From enrollment through 12 months for patients who use PrEP. For the interview only group and clinician group, this information is collected at a single point in time when they are interviewed.
  This outcome measures the proportion of participants who remain on oral PrEP (F/TAF) at 1, 2, 4, 8, and 12 months after initiation in the emergency department. Adherence will be assessed through self-report interviews. Persistence is defined as continued PrEP use without discontinuation during the 12-month follow-up period. This measure will help determine real-world feasibility of maintaining PrEP among persons who use drugs and identify barriers and facilitators to adherence.

SECONDARY OUTCOMES:
Qualitative Themes Related to PrEP Initiation and Continuation | For PrEP using participants: enrollment through 12 months. For interview only and clinician groups: single interview session.
  Themes identified from semi structured interviews examining stigma, access to care, social support, and structural barriers influencing PrEP initiation and continuation among persons who use drugs. Themes will be analyzed using standard qualitative thematic analysis procedures.
Identification and Enrollment of F/TAF Eligible Patients | Enrollment through 12 months.
  Number of patients identified as eligible for F/TAF in the acute care setting and proportion successfully enrolled in the intervention pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Henderson, PhD, MCAP, Principal Investigator — University of South Florida

IPD SHARING:
Plan to Share IPD: No
Information collected as part of the research will not be used or distributed for future research studies.

REFERENCES:
- [Background] World Health Organization (WHO). Guidelines on HIV prevention, diagnosis, treatment and care for key populations. Geneva: WHO; 2016.
- [Background] Taylor SW, Psaros C, Pantalone DW, et al. "Life-Steps" for PrEP adherence: demonstration of a CBT-based intervention to increase adherence to pre-exposure prophylaxis medication among sexual-minority men at high risk for HIV acquisition. Cognitive and Behavioral Practice. 2017;24(1):38-49.
- [Background] Smith DK, Van Handel M, Wolitski RJ. PrEP awareness and attitudes in a national survey of primary care clinicians in the United States, 2009-2015. PLOS ONE. 2020;15(8):e0238372.
- [Background] Sherbuk JE, Kline D, DeHovitz J, Braunstein SL. Linkage to HIV pre-exposure prophylaxis care for people who inject drugs. Journal of the International AIDS Society. 2019;22(S4):e25314.
- [Background] Maryshow TA, Caro J. Pilot study on offering HIV pre-exposure prophylaxis (PrEP) to people who inject drugs (PWID) in the inpatient setting.
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Kunselman AR. A brief overview of pilot studies and their sample size justification. Fertility and Sterility. 2024. https://doi.org/10.1016/j.fertnstert.2024.01.040.
- [Background] Kelley CF, Kahle E, Siegler A, et al. Applying a PrEP continuum of care for people who inject drugs in the United States. Clinical Infectious Diseases. 2020;70(8):1603-1610.
- [Background] Food and Drug Administration (FDA). Descovy® (emtricitabine and tenofovir alafenamide) prescribing information. U.S. Food and Drug Administration.
- [Background] Edelman EJ, Moore BA, Calabrese SK, et al. Primary care physicians' readiness to prescribe HIV pre-exposure prophylaxis for people who inject drugs. Addiction Science & Clinical Practice. 2019;14:35.
- [Background] Choopanya K, Martin M, Suntharasamai P, et al.; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomized, double-blind, placebo-controlled phase 3 trial. Lancet. 2013;381(9883):2083-2090.
- [Background] Centers for Disease Control and Prevention (CDC). U.S. Public Health Service: Preexposure Prophylaxis for the Prevention of HIV Infection in the United States-2021 Update: A Clinical Practice Guideline. Atlanta, GA: CDC; 2021.
- [Background] Biello KB, Bazzi AR, Mimiaga MJ, et al. Perspectives on HIV pre-exposure prophylaxis (PrEP) utilization and related intervention needs among people who inject drugs. Harm Reduction Journal. 2018;15:55. https://doi.org/10.1186/s12954-018-0263-5.
- See also: As described in the Descovy drug pamphlet, pregnancy exposure reporting is standard of care. The study team will register any pregnancies that occur while any female subject is on PrEP to the Antiretroviral Pregnancy Registry (APR) found online. — https://www.apregistry.com/